CLINICAL TRIAL: NCT03097250
Title: MRI Spectroscopy and Neuropsychological Functioning in Phenylketonuria
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Susan Waisbren, Psychologist, Boston Children's Hospital
Other Study IDs: IRB-P00025151
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Phenylketonuria
Keywords: PKU; Neuropsychology; MRI
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PKU Subjects: Subjects with PKU will be asked to undergo an MRI and blood draw on Day 1 and Day 2 of the study. They will also receive neuropsychological testing on Day 1 of the study
- Controls: Controls will undergo only one MRI and blood draw on Day 1 of the study. They will also receive neuropsychological testing on Day 1 of the study.

SUMMARY:
This is a study about the relationship of brain biomarkers with neuropsychological functioning in PKU. All participants will undergo MRI spectroscopy, will provide a blood specimen and will receive neuropsychological testing.

DETAILED DESCRIPTION:
Despite newborn screening and early initiation of treatment, many adolescents and adults with PKU experience some degree of neuropsychological dysfunction or mood disturbances. Blood phenylalanine (Phe) levels and low levels of tyrosine (Tyr) only partially explain why some individuals with PKU have these difficulties and others do not. In this study, the investigators will use a new approach involving magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) for measuring brain Phe (and other brain chemicals) in order to determine relationships between brain biomarkers and neuropsychological functioning and mood. Previously, brain Phe and Tyr could not be reliably measured by MRS methods, especially in concentrations likely to be found in individuals with treated PKU. This project will use an improved method for measuring brain Phe and Tyr. The investigators will use two-dimensional shift correlated magnetic resonance spectroscopy (COSY). COSY is a non-invasive method that allows for quantitative measurement of Phe, Tyr and other amino acids in the brain. This project has the potential to close one of the most important gaps in the knowledge of PKU, namely to define how PKU affects the brain. The aims of this study are to examine brain Phe and Tyr in individuals with PKU and in an age-matched healthy comparison group, and 2) determine the association of Phe and Tyr in distinct brain regions with measures of neuropsychological functioning and mood. Participants with PKU will receive 2 MRI scans with spectroscopy and the comparison group will receive 1 MRI scan with spectroscopy under fasting conditions. All participants will provide a blood specimen for blood amino acid determinations and will receive neuropsychological testing. The investigators will develop statistical models that can be applied in future studies to enhance understanding of PKU. This pilot study is important because it will provide evidence of the usefulness of COSY. COSY has the potential to explain individual differences in PKU, identify specific cognitive functions or mood disturbances related to high brain Phe or low brain Tyr, and offer an additional marker or endpoint for evaluating new treatments in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-25 years
2. Not currently participating in a clinical trial
3. Capable of providing informed assent/consent
4. Able to undergo MRI procedures without sedation
5. Does not have metal implants (braces or permanent retainers made of MRI-compatible materials are permitted since we will not be doing procedures, such as DTI, affected by non-ferrous metals).
6. PKU Group: identified by newborn screening; received treatment within the first 30 days of life
7. PKU Group: Pre-treatment/off-diet blood Phe concentration at or above 600 umol/L

Exclusion Criteria:

1. Older than 25 years or younger than 12 years of age.
2. Currently participating in a clinical trial
3. Incapable of providing informed assent/consent
4. Pregnant women will be excluded
5. Not able to tolerate MRI procedures without sedation
6. Has metal implants or braces on teeth not compatible with MRI
7. Has any known contraindication for MRI
8. PKU Group: Pre-treatment/off-diet blood Phe concentration below 600 umol/L)
9. PKU Group: Not identified through newborn screening or treatment was initiated after 30 days of life

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This is an observational case-controlled study that will include adolescents and young adults with PKU (ages 12-25) and a matched comparison group of healthy individuals of the same age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Neuropsychological functioning | 1 day
  NIH Toolbox Cognitive Battery
Social/Emotional Outcome | 1 day
  NIH PROMIS Questionnaires (Neuro QoL)
Blood Biomarkers | 2 days
  Phenylalanine and Tyrosine (umol/L)
Brain Biomarkers | 2 days
  Phenylalanine and Tyrosine (umol/L)

SECONDARY OUTCOMES:
Intellectual Functioning | 1 day
  Full Scale IQ

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Waisbren, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No